CLINICAL TRIAL: NCT03472703
Title: Effect of Consumption on Cognitive Processes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ERN_10-0014AP7
Record Dates: First submitted 2018-01-17; First posted 2018-03-21 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-03

CONDITIONS: Eating Behavior; Hunger; Inhibition; Functional Magnetic Resonance Imaging
Keywords: fMRI; Cognitive processes; Inhibition; Food reward; Appetite
MeSH Terms: conditions — Feeding Behavior; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: We will use a counter-balanced, crossover, within-subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hungry (Other): Her subjects will first have a break, then undergo all measurement and at the end of the study-day they will receive their lunch
  Interventions: Other: Break-Lunch time
- Satiated (Other): Her subjects will first receive their lunch, then perform all the tasks and last will have a break
  Interventions: Other: Break-Lunch time

INTERVENTIONS:
Other: Break-Lunch time — The time for the break and lunch will be contrary, depending on their visit/session

SUMMARY:
To get a better understanding of the interaction between metabolism, neural responses, cognitive processes and appetite the investigaters will examine the effect of food consumption on cognitive processes. The investigaters will look at the effect of satiation on cognitive performance on both a behavioural and neuronal level. In this study participants will undergo functional magnetic resonance imaging (fMRI) measurements while performing a food reward and inhibition task, and in addition perform a memory, working memory and delay discount task, once when hungry and once when full.

DETAILED DESCRIPTION:
Human eating behaviour is a very complex process. It has been well established that food intake and choice are influences by nutritional composition of the food and their reward values. However recent work suggests that cognitive processes such as memory, attention, and inhibition influence food choices. Thinking about food can lead to increased attention to food cues, which can result in a greater chance of actual food consumption. Additional manipulation of attention effects memory and snack intake. It has been suggested that memory inhibition plays a critical role in suppression of food-related information when satiated to prevent overeating. These results underpin the interaction between cognitive processes and internal state and its effect on appetite. Although it has been widely studied what the effect of satiation is on reward and even which brain regions are associated with food intake, for both homeostatic and hedonic eating, the direct effect of consumption on cognitive processes and the related brain processes are rather unknown.

In this study participants will be asked to come to a research facility twice (within-design). Once the particpant will undergo all the tasks when hungry and receive a lunch at the end of the study-day (hungry session), and once the subject will first receive a lunch and then perform all the tasks (satiated session). Upon arrival subjects will fill in their appetite and mood ratings, followed by a break or a lunch (depending on the session). After the 25-min break/lunch the subject will be placed in the scanner. First the particpants neural responses will be measure while performing an inhibition task, here subjects will complete a go-no/go task; the particpant either has to go (press) when seeing a toiletry or stationary item, or not go (withhold pressing) when seeing a food or sports item. Second a resting state fMRI measurement will be performed. Third subjects will see food and non-food items, which the particpant has to rate on their appeal. Last an anatomical scan will be run. When out of the scanner subjects will undergo several cognitive computerized tasks, a word recall task, a working memory task (measuring the top-down guidance of attention to food stimuli via working memory) and a delay discount task. At last subjects will get lunch (when receiving a break at the start) or a break (when consuming food at arrival).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age 18-45 years at start of the study
* Right-handedness (including left-handers could bias the results because of the laterality of brain functions)
* Ability to give informed consent
* Fluent English speaking
* Willingness to be informed about chance findings of pathology

Exclusion Criteria:

* Subjects who have a non-removable metal object in or at their body, such as, for example: Heart pace-maker, artificial heart valve, metal prosthesis, implants or splinters, non-removable dental braces
* Tattoos, that are older than 15 years
* Claustrophobia
* Pathological hearing ability or an increased sensitivity to loud noises
* Lack of ability to give informed consent
* Operation less than three months ago
* Acute illness or infection during the last 4 weeks
* Cardiovascular disorders (e.g., hypertrophic cardiomyopathy, long QT syndrome)
* Moderate or severe head injury
* Eating disorders
* No metabolic (e.g. metabolic disorder, diabetes, insulin resistance), psychological (e.g. depression) or neurological (e.g. epilepsy, headache disorder, multiple sclerosis, traumatic brain injuries) diseases or medication in relation to these diseases.
* Current weight loss regimens, or more then 5kg weight loss in the last 3 months
* Smoking
* Current pregnancy or breastfeeding
* Current or past history of drug or alcohol dependency - alcohol consumption exceeding 12 units a week
* Food allergies (e.g. peanut allergy lactose and gluten intolerance) or vegetarian/vegan diet
* Disliking the study lunch

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
fMRI brain responses during inhibition | 14 minutes
  - Neural activation correct No-Go vs. Go trail. Subjects neural activation when they are instructed to go (press) when seeing toiletry or stationary items and react correctly compared to when subjects are instructed not to go (no press) when seeing a food or sport and withhold correctly
fMRI brain repsonse during inhibition to a food stimuli | 14 minutes
  Neural activation during correct inhibition food vs. non-food stimuli trail. Comparing the brain response when subjects correctly withhold for food vs a sports item.
fMRI neural network during inhibition to a food stimuli | 14 minutes
  Functional connectivity during correct inhibition food vs. non-food stimuli trail.

SECONDARY OUTCOMES:
Word recall | 10 minutes
  Recall accuracy. The researchers will count the correct amount of words remembered in this task and calculate % of words remembered in total, and differentiate between the three categories (food/neutral/emotional)
Delay discount of food reward | 10 minutes
  - Area under the curve for delay of choosing a food item. Subjects have to choice between a certain amount of food now, or more (which varies between 1-20 pieces) food later (which will vary from 1 day, 1 months and 1 year).
Delay discount of money reward | 10 minutes
  - Area under the curve for delay of choosing a amount of money. Subjects have to choice between a certain amount of money now, or more (which varies between 1-100 pound) money later (which will vary from 1 day, 1 months and 1 year).
Reaction time to target | 25 minutes
  Particpants have to hold a food or non-food image in working memory for later retrieval. Subsequently, particpants have to respond to a target and ignore a distracter, both paired with an image. As a outcome there are three reaction time critical conditions (i) valid trials, when the memorized item appeared next to the search target; (ii) invalid trials, when the memorized item appeared next to a distracter in the search display; (iii) neutral trials in which the memorized item did not re-appear in the search display. The
fMRI brain activity in food picture task | 18 minutes
  - Brain responses for food stimuli compared to non-food stimuli. We will measure this by showing subjects food and non-food images while preforming and fMRI-scan and subtract activity during non-food images from the activity pattern when looking at food images.

CONTACTS AND LOCATIONS:
Overall Officials: Maartje S Spetter, PhD, Principal Investigator — UoB
Locations (1):
- University of Birmingham School of Psychology, Birmingham, Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided